CLINICAL TRIAL: NCT02182362
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of 20 mg, 48 mg, 120 mg, and 240 mg Once a Day of BI 201335 NA (Oral Solution) in Healthy Male Subjects, in a Randomized Double Blind, Placebo Controlled Study
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Doses of BI 201335 NA in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.6
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- BI 201335 NA in rising doses (Experimental): single dose of BI 201335 NA on day 1, multiple dosing days 4-24
  Interventions: Drug: BI 201335 NA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 201335 NA (Experimental): highest tolerated dose of BI 201335 on day 1-28 in patients with Gilbert's syndrome
  Interventions: Drug: BI 201335 NA

INTERVENTIONS:
Drug: BI 201335 NA
  Arms: BI 201335 NA; BI 201335 NA in rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main objective was to investigate the safety, tolerability and the pharmacokinetics (PK) of BI 201335 NA in healthy male subjects without Gilbert's syndrome or polymorphism (GS) following oral administration of a single dose (Day 1) and repeated doses (Days 4-24) of 20 mg, 48 mg, 120 mg, and 240 mg. Additionally, the safety, tolerability, and the PK of the highest tolerated dose of BI 201335 NA (determined during the multiple-rising-dose phase) were assessed in healthy male subjects with GS over a 28-day continuous drug administration period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria:

  * Complete medical history, physical examination, vital signs (Blood Pressure, Pulse Rate), 12-lead ECG (electrocardiogram), and clinical laboratory tests
* Age ≥18 and Age ≤55 years
* BMI ≥18.5 and BMI ≤30 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Subjects with polymorphisms associated with Gilbert's syndrome will be excluded from the initial 4 groups of the multiple rising dose phase of the study. However, only subjects with Gilbert's polymorphism will be allowed to participate in the last group which will be treated with the highest tolerated dose determined in the multiple rising dose phase of the trial
* Prior history of jaundice for subjects without Gilbert's polymorphism
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 30 days prior to screening until trial completion
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoking (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during the trial
* Alcohol abuse (more than 60 g/day)
* Inability to refrain from alcohol during the trial
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for TdP (Torsades de points) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline and up to 46 days
Number of patients with clinically relevant changes in vital signs (blood pressure (BP), pulse rate (PR)) | Baseline and up to 32 days
Number of patients with clinically relevant changes in 12-lead ECG (electrocardiogram) | Baseline and up to 32 days
Number of patients with clinically relevant changes in clinical laboratory tests (haematology, clinical chemistry, urinalysis) | Baseline and up to 32 days
Incidence of adverse events | up to day 46
Assessment of tolerability by investigator | Day 28 or 32

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
λz (terminal rate constant in plasma) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
t1/2 (terminal half-life of the analyte in plasma) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
MRTpo (mean residence time of the analyte in the body after single oral administration) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
CL/F (apparent clearance of the analyte in plasma) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
Vz/F (apparent volume of distribution during the terminal phase λz) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60 hours after first treatment
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
λz,ss (terminal rate constant in plasma at steady state) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
CL/F,ss (apparent clearance of the analyte in the plasma at steady state following multiple oral dose administration) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following oral administration) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours after last dose